CLINICAL TRIAL: NCT00005219
Title: Predicting Physical Activity Change: an Epidemiologic Study
Status: Completed | Type: Observational
Sponsor: San Diego State University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Melbourne Hovell, Professor, San Diego State University
Other Study IDs: 1098; R01HL040575 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Exercise Study Participants: Data from the San Diego Health and Exercise Baseline survey conducted in 1986 were used to contact participants for the follow-up

SUMMARY:
To conduct a two-year follow up of participants in a cross-sectional study of physical activity determinants. Predictors of change in vigorous exercise habits and recreational walking habits were identified as were determinants of change in the proportion of the sample who initiated, maintained, or discontinued exercise.

DETAILED DESCRIPTION:
BACKGROUND:

In 1988 when the study began, epidemiological studies had shown the health benefits of physical activity and that prevalence of physical activity was well below recommended levels. Exercise-promotion interventions were typically ineffective, and lack of knowledge of exercise determinants inhibited the design of effective interventions.

DESIGN NARRATIVE:

Data from the San Diego Health and Exercise Baseline survey conducted in 1986 were used to contact participants for the follow-up. The difference in reported activity level from time 1 to time 2 served as an estimate of change in activity. The follow-up survey elicited a two-year history of vigorous exercise and moderate-intensity exercise, both of which have substantial health benefits, as well as different determinants. Potential predictors were assessed at baseline and included demographic variables and indices based on social learning theory. Multiple regression analyses determine the combined and independent relationships of such variables as self-efficacy, social support, perceived barriers and benefits and environmental factors on both types of physical activity change. A second analysis separated subjects into the baseline physical activity groups of low, intermediate, and high activity and examined prediction of change versus no-change in each category.

ELIGIBILITY:
Inclusion

1. Healthy Adults 18-60

   Exclusion
2. Cardiovascular Disease
3. Heart Disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Healthy Adults 18-60
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 1988-04 (Actual); Primary Completion 1990-04 (Actual); Study Completion 1991-04 (Actual)

PRIMARY OUTCOMES:
Minutes of exercise | Over 2 years
  Change in minutes of exercise from pre to post

CONTACTS AND LOCATIONS:
Overall Officials: J F Sallis, Study Director — San Diego State University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hovell MF, Hofstetter CR, Sallis JF, Rauh MJ, Barrington E. Correlates of change in walking for exercise: an exploratory analysis. Res Q Exerc Sport. 1992 Dec;63(4):425-34. doi: 10.1080/02701367.1992.10608765. PMID 1439168
- [Background] Hofstetter CR, Sallis JF, Hovell MF. Some health dimensions of self-efficacy: analysis of theoretical specificity. Soc Sci Med. 1990;31(9):1051-6. doi: 10.1016/0277-9536(90)90118-c. PMID 2255964
- [Background] Sallis JF, Hovell MF. Determinants of exercise behavior. Exerc Sport Sci Rev. 1990;18:307-30. No abstract available. PMID 2192898
- [Background] Sallis JF, Hovell MF, Hofstetter CR. Predictors of adoption and maintenance of vigorous physical activity in men and women. Prev Med. 1992 Mar;21(2):237-51. doi: 10.1016/0091-7435(92)90022-a. PMID 1579558
- [Background] Sallis JF, Hovell MF, Hofstetter CR, Barrington E. Explanation of vigorous physical activity during two years using social learning variables. Soc Sci Med. 1992 Jan;34(1):25-32. doi: 10.1016/0277-9536(92)90063-v. PMID 1738853
- [Background] Sallis JF, Hovell MF, Hofstetter CR, Elder JP, Faucher P, Spry VM, Barrington E, Hackley M. Lifetime history of relapse from exercise. Addict Behav. 1990;15(6):573-9. doi: 10.1016/0306-4603(90)90059-7. PMID 2075855